CLINICAL TRIAL: NCT02699099
Title: Immunogenicity and Safety Study of GSK Biologicals' Candidate Malaria Vaccine (SB257049) Given at 6, 7.5 and 9 Months of Age in Co-administration With Measles, Rubella and Yellow Fever Vaccines Followed by a Booster of the Malaria Vaccine.
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Candidate Malaria Vaccine Given at 6, 7.5 and 9 Months of Age in Co-administration With Measles, Rubella and Yellow Fever (YF) Vaccines Followed by a Booster of the Malaria Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200596
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Children; Infants; SB257049; Malaria; Immunogenicity; Surveillance; Efficacy; Safety; Africa; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Vitamin A; RTS malaria vaccine; Rubella Vaccine; Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coad group (Experimental): Children randomized received Vitamin A at 6 months of age, SB257049 vaccine at 6, 7.5 and 9 months of age, and Yellow Fever (YF) vaccine and a combined measles and rubella vaccine at 9 months of age. Subjects received a booster dose of SB257049 vaccine at 18 months post Dose 3 (i.e. at 27 months of age).
  Interventions: Dietary Supplement: Vitamin A; Biological: Candidate Plasmodium falciparum malaria vaccine; Biological: MR-Vac; Biological: Stamaril
- RTS,S group (Experimental): Children randomized received Vitamin A at 6 months of age, SB257049 vaccine at 6, 7.5 and 9 months of age, and Yellow Fever (YF) vaccine and a combined measles and rubella vaccine at 10.5 months of age. Subjects received a booster dose of SB257049 vaccine at 18 months post Dose 3 (i.e. at 27 months of age).
  Interventions: Dietary Supplement: Vitamin A; Biological: Candidate Plasmodium falciparum malaria vaccine; Biological: MR-Vac; Biological: Stamaril
- Control group (Experimental): Children randomized received Vitamin A at 6 months of age and Yellow Fever (YF) vaccine and a combined measles and rubella vaccine at 9 months of age. These children received SB257049 vaccine at 10.5, 11.5 and 12.5 months of age plus a booster dose 17.5 months post Dose 3 (i.e. at 30 months of age).
  Interventions: Dietary Supplement: Vitamin A; Biological: Candidate Plasmodium falciparum malaria vaccine; Biological: MR-Vac; Biological: Stamaril

INTERVENTIONS:
Dietary Supplement: Vitamin A — Oral administration of Vitamin A (1 dose)
Biological: Candidate Plasmodium falciparum malaria vaccine — Intramuscular administration of SB257049 vaccine (4 doses)
  Other Names: GSK Biologicals' candidate Plasmodium falciparum malaria vaccine adjuvanted with GSK Biologicals' proprietary Adjuvant System AS01E (RTS,S/AS01E)
Biological: MR-Vac — Subcutaneous injection of a combined measles and rubella vaccine (1 dose)
  Other Names: Live attenuated measles virus and rubella virus vaccine (MR-Vac)
Biological: Stamaril — Intramuscular injection of a yellow fever (YF) vaccine (1 dose)
  Other Names: Yellow Fever (YF) Vaccine

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety, and reactogenicity of the SB257049 candidate malaria vaccine when co-administered with Vitamin A, measles, rubella and yellow fever vaccines to children aged 6 months at the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) (LAR[s]) who, in the opinion of the investigator, could and complied with the requirements of the protocol.
* A male or female 6 months of age (from the day the child becomes 6 months of age until the day before the child achieved 7 months of age) at the time of the first vaccination.
* Signed or thumb-printed informed consent obtained from the parent(s)/LAR(s) of the subject. Where parent(s)/LAR(s) were illiterate, the consent form was countersigned by an independent witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously received three documented doses of diphtheria, tetanus, and whole-cell pertussis, hepatitis B vaccine (DTPwHepB), and a 3-dose course of oral polio vaccine and, if locally recommended, pneumococcal and rotavirus vaccines.

Exclusion Criteria:

* Child in care
* Use of a drug or vaccine that is not approved for that indication other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this meant prednisone≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids were allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting seven days before the first dose of SB257049 measles, rubella and YF vaccines and ending 42 days after the last dose of vaccines given at 9 months of age (Visit 4), with the exception of oral polio vaccine which could be given for unforeseen public health threat.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination against measles, YF or rubella.
* Previous administration of Vitamin A.
* Moderate or severe malnutrition at screening defined as weight for age Z-score < -2.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s). See also Section 1.3.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment. Fever was defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route for recording temperature in this study was axillary.

Subjects with a minor illness without fever might have been enrolled at the discretion of the investigator.

* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Same sex twin.
* Maternal death.
* Previous participation in any other malaria study.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 699 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Kumasi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coad Group | RTS,S Group | Control Group
Started | 231 | 236 | 232
Completed | 223 | 233 | 226
Not Completed | 8 | 3 | 6
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 7 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coad Group | RTS,S Group | Control Group | Total
Number analyzed (Participants) | 231 | 236 | 232 | 699
Age, Continuous [Mean (Standard Deviation); unit: Months] | 6.3 (0.3) | 6.3 (0.3) | 6.3 (0.3) | 6.3 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 119 | 113 | 348
  Male | 115 | 117 | 119 | 351
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 231 | 236 | 232 | 699

OUTCOME MEASURES:

1. Primary Outcome: Anti-Circumsporozoite (Anti-CS) Antibody Concentrations, One Month Post Dose 3 of SB257049 (Primary Analysis)
Description: Concentrations were expressed as Geometric Mean Concentrations (GMCs) with the following unit of measure: Enzyme Linked Immunosorbent Assay (ELISA) units per milliliter (EU/mL). The 95% confidence intervals were calculated using the Analysis of Variance (ANOVA) model. The antibody response of anti-CS was assessed in the Coad Group and the RTS,S Group.
Time Frame: At one month post Dose 3 of SB257049 (Month 4)
Population: Analysis was performed on the Per-Protocol set for immunogenicity defined for the primary analysis (Month 4.5), which included all evaluable subjects meeting all eligibility criteria, complying with protocol defined procedures, with no elimination criteria during the study. Subjects with incomplete vaccination course or blood sampling outside protocol windows were eliminated.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 207 | 213
EU/mL | 452.87 [409.85 to 500.41] | 422.49 [382.89 to 466.18]
Statistical Analysis 1: Comparison: Coad Group vs RTS,S Group; Adjusted GMC ratios for anti-CS antibody: To demonstrate the non-inferiority of the antibody response to the CS antigen when SB257049 is co-administered with YF vaccine and a combined measles and rubella vaccine versus SB257049 administered alone; Test type: Non-Inferiority — Non-inferiority (1 month post-Dose 3 of SB257049) was defined as the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio (RTS,S group/Coad group) for anti-CS, being below a limit of 2; ANOVA; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]

2. Secondary Outcome: Anti-CS Antibody Concentrations, Pre-vaccination and One Month Post Dose 3 of SB257049
Description: Concentrations were expressed as Geometric Mean Concentrations (GMCs) with the following unit of measure: ELISA units per milliliter (EU/mL). The 95% CI for the GMC was obtained by exponential transformation (base 10) of the 95% CI for the mean of the log transformed concentrations. The antibody response of anti-CS was assessed in the Coad Group and the RTS,S Group.
Time Frame: At Day 0 and one month post Dose 3 of SB257049 (Month 4)
Population: Analysis was performed on the Per-Protocol set for immunogenicity, defined at study end, which included all evaluable subjects meeting all eligibility criteria, complying with protocol defined procedures, with no elimination criteria during the study. Subjects with incomplete vaccination course or blood sampling performed outside protocol defined windows were eliminated.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 208 | 213
EU/mL
  Anti-CS - Day 0 | 0.96 [0.94 to 0.97] | 0.96 [0.94 to 0.98]
  Anti-CS - Month 4 | 454.51 [408.58 to 505.60] | 422.49 [385.42 to 463.12]

3. Secondary Outcome: Number of Seropositive Subjects for Anti-CS Antibodies, Pre-vaccination and One Month Post Dose 3 of SB257049
Description: A subject seropositive for anti-CS antibody was a subject whose antibody concentration was greater than or equal (≥) to the cut-off value (anti-CS ≥ 1.9 ELISA unit per milliliter [EU/mL]). Seropositivity was assessed in the Coad Group and the RTS,S Group.
Time Frame: At Day 0 and one month post Dose 3 of SB257049 (Month 4)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 208 | 213
Participants
  Anti-CS - Day 0 | 1 | 2
  Anti-CS - Month 4 | 207 | 213

4. Secondary Outcome: Anti-hepatitis B (Anti-HBs) Antibody Concentrations, Pre-vaccination and One Month Post-Dose 3 of SB257049
Description: Concentrations were expressed as GMCs with the following unit of measure: milli-international unit per milliliter (mIU/mL). The antibody response of anti-HB was assessed in the Coad Group and the RTS,S Group.
Time Frame: At Day 0 and one month post Dose 3 of SB257049 (Month 4)
Population: Analysis was performed on the Per-Protocol set for immunogenicity which included all evaluable subjects meeting all eligibility criteria, complying with protocol defined procedures, with no elimination criteria during the study, and who had available data concerning the outcome measure. Subjects with incomplete vaccination course or blood sampling performed outside protocol defined windows were eliminated.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 205 | 210
mIU/mL
  Anti-HBs - Day 0: number analyzed (Participants) | 205 | 208
  Anti-HBs - Day 0 | 397.36 [318.21 to 496.18] | 427.65 [340.47 to 537.14]
  Anti-HBs - Month 4 | 42162.55 [35643.11 to 49874.45] | 43261.19 [37275.19 to 50208.47]

5. Secondary Outcome: Number of Seroprotected Subjects for Anti-HB Antibodies, Pre-vaccination and One Month Post-Dose 3 of SB257049
Description: Seroprotection rate for anti-HBs antibody was defined as the percentage of subjects with antibody concentrations greater than or equal to an established cut-off value (anti-HBs ≥ 10 milli-international unit per milliliter [mIU/mL]). Seroprotection was assessed in the Coad Group and the RTS,S Group.
Time Frame: At Day 0 and one month post-Dose 3 of SB257049 (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 205 | 210
Participants
  Anti-HB - Day 0: number analyzed (Participants) | 205 | 208
  Anti-HB - Day 0 | 196 | 201
  Anti-HB - Month 4 | 205 | 210

6. Secondary Outcome: Number of Seroconverted Subjects for Anti-Measles (Anti-Me) Antibodies, One Month Post-vaccination With the Combined Measles and Rubella (MeRu) Vaccine
Description: Seroconversion was defined as number of subjects with an anti-Measles antibodies pre-vaccination concentration below 150 mIU/mL and a post-vaccination concentration ≥150 mIU/mL. Seroconversion was assessed in the Coad group and the Control group.
Time Frame: At one month post-vaccination with the combined measles and rubella (MeRu) vaccine (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 205 | 216
Participants | 197 | 212
Statistical Analysis 1: Comparison: Coad Group vs Control Group; Difference in seroconversion rates against measles antibodies: To demonstrate the non-inferiority of the antibody response to the measles vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered with SB257049 versus administration without SB257049; Test type: Non-Inferiority — Non-inferiority was defined as the upper limit of the 95% confidence interval (CI) for the difference in seroconversion rate of the anti-measles antibody, being below 10% for the two groups (Control Group minus Coad Group); Miettinen and Nurminen method; Miettinen and Nurminen method was used to construct 95%CI for difference between groups; Difference in percentage = 2.05, 95% CI 2-sided [-1.29 to 5.89]

7. Secondary Outcome: Anti-Me Antibody Concentrations, Pre-vaccination and One Month Post-vaccination With the Combined Measles and Rubella Vaccine
Description: Concentrations were expressed in GMCs with the following unit of measure: milli-international unit per milliliter (mIU/mL). The antibody response of anti-Me was assessed in the Coad Group and the Control Group.
Time Frame: At pre-vaccination (Month 3) and one month post-vaccination with combined measles and rubella vaccine (Month 4)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 208 | 220
mIU/mL
  Anti-Me - Month 3: number analyzed (Participants) | 205 | 220
  Anti-Me - Month 3 | 75.00 [75.00 to 75.00] | 75.00 [75.00 to 75.00]
  Anti-Me - Month 4: number analyzed (Participants) | 208 | 217
  Anti-Me - Month 4 | 565.81 [513.40 to 623.57] | 572.09 [523.83 to 624.79]

8. Secondary Outcome: Number of Seropositive Subjects for Anti-Me Antibodies, Pre-vaccination and One Month Post-vaccination With the Combined Measles and Rubella Vaccine
Description: A subject seropositive for anti-CS antibody was a subject whose antibody concentration was greater than or equal (≥) to the cut-off value (anti-Me ≥ 150 mIU/mL). Seropositivity was assessed in the Coad Group and the Control Group.
Time Frame: At pre-vaccination (Month 3) and one month post-vaccination with the combined measles and rubella vaccine (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 208 | 220
Participants
  Anti-Me - Month 3: number analyzed (Participants) | 205 | 220
  Anti-Me - Month 3 | 0 | 0
  Anti-Me - Month 4: number analyzed (Participants) | 208 | 217
  Anti-Me - Month 4 | 200 | 213

9. Secondary Outcome: Number of Seroconverted Subjects for Anti-Rubella (Anti-Ru) Antibodies, One Month Post-vaccination With the Combined Measles and Rubella Vaccine
Description: Seroconversion was defined as number of subjects with an anti-Ru pre-vaccination concentration less than (<) 4 IU/mL and a post-vaccination concentration ≥ 4 IU/mL. Seroconversion was assessed in the Coad group and Control group.
Time Frame: At one month post-vaccination with combined measles and rubella vaccine (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 200 | 212
Participants | 199 | 212
Statistical Analysis 1: Comparison: Coad Group vs Control Group; Difference in seroconversion rates against Rubella antibodies: To demonstrate the non-inferiority of the antibody response to the rubella vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered. with SB257049 versus administration without SB257049; Test type: Non-Inferiority — Non-inferiority was defined as the upper limit of the 95% confidence interval (CI) for the difference in seroconversion rates of the anti-rubella antibody, being below 10% for the two groups (Control Group minus Coad Group); Miettinen and Nurminen method; Miettinen and Nurminen method was used to construct 95%CI for difference between groups; Difference in percentage = 0.50, 95% CI 2-sided [-1.29 to 2.78]

10. Secondary Outcome: Anti-Ru Antibody Concentrations, Pre-vaccination and One Month Post-vaccination With the Combined Measles and Rubella Vaccine
Description: Concentrations were expressed as GMCs with the following unit of measure: International unit per milliliter (IU/mL). The antibody response of anti-Ru was assessed in the Coad Group and Control Group.
Time Frame: At pre-vaccination (Month 3) and one month post-vaccination with combined measles and rubella vaccine (Month 4)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 208 | 220
IU/mL
  Anti-Ru - Month 3: number analyzed (Participants) | 205 | 220
  Anti-Ru - Month 3 | 2.08 [1.99 to 2.18] | 2.09 [1.98 to 2.20]
  Anti-Ru - Month 4: number analyzed (Participants) | 208 | 217
  Anti-Ru - Month 4 | 39.36 [35.20 to 44.01] | 42.45 [38.42 to 46.92]

11. Secondary Outcome: Number of Seropositive Subjects for Anti-Ru Antibodies, Pre-vaccination and One Month Post-vaccination With the Combined Measles and Rubella Vaccine
Description: A subject seropositive for anti-Ru antibody was a subject whose antibody concentration was greater than or equal (≥) to the cut-off value (anti-Ru ≥ 4 IU/mL). Seropositivity was assessed in the Coad Group and Control Group.
Time Frame: At pre-vaccination (Month 3) and one month post-vaccination with combined measles and rubella vaccine (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 208 | 220
Participants
  Anti-Ru - Month 3: number analyzed (Participants) | 205 | 220
  Anti-Ru - Month 3 | 5 | 4
  Anti-Ru - Month 4: number analyzed (Participants) | 208 | 217
  Anti-Ru - Month 4 | 207 | 217

12. Secondary Outcome: Number of Seropositive Subjects for Anti-Yellow Fever (Anti-YF) Antibodies, at One Month Post-vaccination With the YF Vaccine
Description: Seropositivity was defined as number of subjects with anti-YF titers greater than or equal to (≥) 10 End point Dilution 50 (ED50). Seropositivity was assessed in the Coad group and Control group.
Time Frame: At one month post-vaccination with the YF vaccine (Month 4)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 207 | 217
Participants | 203 | 214
Statistical Analysis 1: Comparison: Coad Group vs Control Group; Difference in seropositivity rates against Yellow Fever antibodies: To demonstrate the non-inferiority of the antibody response to the YF vaccine antigen when YF vaccine and a combined measles and rubella vaccine are coadministered with SB257049 versus administration without SB257049; Test type: Non-Inferiority — Non-inferiority was defined as the upper limit of the 95% confidence interval (CI) for the difference in seropositivity rates of the anti-yellow fever antibody , being below 10% for the two groups (Control Group minus Coad Group); Miettinen and Nurminen method; Miettinen and Nurminen method was used to construct 95%CI for difference between groups; Difference in percentage = 0.55, 95% CI 2-sided [-2.30 to 3.65]

13. Secondary Outcome: Anti-YF Antibody Titers One Month Post-vaccination With the YF Vaccine
Description: Titers were expressed as Geometric Mean Titres (GMTs). The antibody response of anti-YF was assessed in the Coad Group and Control Group.
Time Frame: At one month post-vaccination with the YF vaccine (Month 4)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Coad Group | Control Group
Number analyzed (Participants) | 207 | 217
Titers | 324.31 [273.54 to 384.51] | 346.60 [296.73 to 404.86]

14. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms for Coad Group and RTS,S Group After Administration of Vitamin A and Study Vaccines at 6 Months of Age
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = subject crying when limb was moved /spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) at injection site.
Time Frame: During a 7-day follow-up period (day of administration and 6 subsequent days) after administration of Vitamin A and SB257049 dose 1 (Day 0)
Population: Analysis was performed on the Exposed set which included all subjects with the first dose of SB257049 and Vitamin A administered (Coad and RTS,S Groups).
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 231 | 236
Participants
  Pain - Any | 25 | 16
  Pain - Grade 3 | 0 | 1
  Redness - Any | 7 | 13
  Redness - Grade 3 | 0 | 0
  Swelling - Any | 8 | 6
  Swelling - Grade 3 | 0 | 0

15. Secondary Outcome: Number of Subjects With Any, Grade 3, Related, Grade 3 and Related Solicited General Symptoms for the Coad Group and RTS,S Group After Administration of Vitamin A and Study Vaccines at 6 Months of Age
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness, loss of appetite, measles/rubella-like rash and fever. Any = occurrence of the symptom regardless of intensity grade. Any Fever = temperature greater than or equal to (≥) 37.5° C (axillary route). Grade 3 drowsiness= symptom that prevented normal activity; Grade 3 Irritability/Fussiness = Crying that couldn't be comforted/prevented normal activity; Grade 3 Loss of appetite = not eating at all; Grade 3 Measles /rubella rash = >150 lesions; Grade 3 fever= temperature grater than (>) 39°C; Related = symptom assessed by the investigator as causally related to the vaccination.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 231 | 235
Participants
  Drowsiness - Any | 4 | 4
  Drowsiness - Grade 3 | 0 | 0
  Drowsiness - Related | 0 | 0
  Drowsiness - Grade 3 related | 0 | 0
  Irritability/Fussiness - Any | 14 | 22
  Irritability/Fussiness - Grade 3 | 1 | 1
  Irritability/Fussiness - Related | 2 | 1
  Irritability/Fussiness - Grade 3 related | 0 | 0
  Loss of appetite - Any | 5 | 7
  Loss of appetite - Grade 3 | 0 | 0
  Loss of appetite - Related | 0 | 0
  Loss of appetite - Grade 3 related | 0 | 0
  Measles/Rubella-like rash - Any | 0 | 0
  Measles/Rubella-like rash - Grade 3 | 0 | 0
  Measles/Rubella-like rash - Related | 0 | 0
  Measles/Rubella-like rash - Grade 3 related | 0 | 0
  Fever - Any | 32 | 30
  Fever - Grade 3 | 3 | 1
  Fever - Related | 10 | 8
  Fever - Grade 3 related | 1 | 0

16. Secondary Outcome: Number of Subjects With Any, Grade 3, Related, Grade 3 and Related Solicited General Symptoms for the Control Group After Administration of Vitamin A at 6 Months of Age
Description: as for outcome 15
Time Frame: During a 7-day follow-up period (day of administration and 6 subsequent days) after administration of Vitamin A (Day 0)
Population: Analysis was performed on the Exposed set which included all subjects with Vitamin A administered (Control group). In the Control Group, only solicited general symptoms were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 232
Participants
  Drowsiness - Any | 1
  Drowsiness - Grade 3 | 0
  Drowsiness - Related | 0
  Drowsiness - Grade 3 related | 0
  Irritability/Fussiness - Any | 6
  Irritability/Fussiness - Grade 3 | 1
  Irritability/Fussiness - Related | 0
  Irritability/Fussiness - Grade 3 related | 0
  Loss of appetite - Any | 9
  Loss of appetite- Grade 3 | 0
  Loss of appetite- Related | 0
  Loss of appetite- Grade 3 related | 0
  Measles/Rubella-like rash - Any | 0
  Measles/Rubella-like rash - Grade 3 | 0
  Measles/Rubella-like rash - Related | 0
  Measles/Rubella-like rash - Grade 3 related | 0
  Fever - Any | 11
  Fever - Grade 3 | 0
  Fever - Related | 1
  Fever - Grade 3 related | 0

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms for Coad Group and RTS,S Group After Dose of Study Vaccines Administered at 7.5 Months of Age
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = subject crying when limb was moved /spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimetres (mm) at injection site.
Time Frame: During a 7-day follow-up period (day of administration and 6 subsequent days) after administration of SB257049 dose 2 (Month 1.5)
Population: Analysis was performed on the Exposed set which included all subjects with the second dose of SB257049 administered (Coad and RTS,S Groups).
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 224 | 234
Participants
  Pain - Any | 3 | 12
  Pain - Grade 3 | 0 | 0
  Redness - Any | 4 | 2
  Redness - Grade 3 | 1 | 0
  Swelling - Any | 4 | 6
  Swelling - Grade 3 | 0 | 0

18. Secondary Outcome: Number of Subjects With Any, Grade 3, Related, Grade 3 and Related Solicited General Symptoms for the Coad Group and RTS,S Group After Dose of Study Vaccines Administered at 7.5 Months of Age
Description: as for outcome 15
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 224 | 234
Participants
  Drowsiness - Any | 6 | 5
  Drowsiness - Grade 3 | 0 | 0
  Drowsiness - Related | 1 | 2
  Drowsiness - Grade 3 related | 0 | 0
  Irritability/Fussiness - Any | 11 | 13
  Irritability/Fussiness - Grade 3 | 0 | 1
  Irritability/Fussiness - Related | 4 | 2
  Irritability/Fussiness - Grade 3 related | 0 | 0
  Loss of appetite - Any | 6 | 11
  Loss of appetite - Grade 3 | 0 | 0
  Loss of appetite - Related | 1 | 0
  Loss of appetite - Grade 3 related | 0 | 0
  Measles/Rubella-like rash - Any | 0 | 0
  Measles/Rubella-like rash - Grade 3 | 0 | 0
  Measles/Rubella-like rash - Related | 0 | 0
  Measles/Rubella-like rash - Grade 3 related | 0 | 0
  Fever - Any | 47 | 47
  Fever - Grade 3 | 3 | 3
  Fever - Related | 11 | 9
  Fever - Grade 3 related | 1 | 1

19. Secondary Outcome: Number of Subjects With Solicited General Symptoms for the Control Group, After Visit at 7.5 Months of Age
Description: Solicited symptoms were not analyzed for the Control Group after visit at Month 1.5 because no vaccination was administered at that visit.
Time Frame: After visit at Month 1.5
Population: Analysis was not performed. Solicited symptoms were not collected for the Control group after visit at Month 1.5 because no vaccination was administered.
Arm/Group | Control Group
Number analyzed (Participants) | 0

20. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms for All Groups, After Dose of Study Vaccines Administered at 9 Months of Age
Description: as for outcome 14
Time Frame: During a 14-day follow-up period (day of administration and 13 subsequent days) after administration of SB257049 dose 3 in Coad (and MeRu+YF) and RTS,S Groups and after MeRu+YF vaccines in Control Group (Month 3)
Population: Analysis was performed on the Exposed set which included all subjects with SB257049 dose 3 for Coad (and MeRu+YF vaccines) and RTS,S Groups, and MeRU+YF vaccines for Control Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 221 | 228 | 225
Participants
  Pain - Any | 10 | 10 | 1
  Pain - Grade 3 | 0 | 0 | 0
  Redness - Any | 0 | 1 | 2
  Redness - Grade 3 | 0 | 0 | 0
  Swelling - Any | 3 | 3 | 1
  Swelling - Grade 3 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Any, Grade 3, Related, Grade 3 and Related Solicited General Symptoms for All Groups, After Dose of Study Vaccines Administered at 9 Months of Age
Description: as for outcome 15
Time Frame: as for outcome 20
Population: Analysis was performed on the Exposed set which included all subjects with SB257049 dose 3 for Coad (and MeRu + YF vaccines) and RTS,S Groups, and MeRU+YF vaccines for Control Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 221 | 229 | 225
Participants
  Drowsiness - Any | 7 | 6 | 0
  Drowsiness - Grade 3 | 0 | 0 | 0
  Drowsiness - Related | 4 | 5 | 0
  Drowsiness - Grade 3 related | 0 | 0 | 0
  Irritability/Fussiness - Any | 11 | 8 | 1
  Irritability/Fussiness - Grade 3 | 0 | 0 | 0
  Irritability/Fussiness - Related | 4 | 4 | 0
  Irritability/Fussiness - Grade 3 related | 0 | 0 | 0
  Loss of appetite - Any | 8 | 6 | 2
  Loss of appetite - Grade 3 | 0 | 0 | 0
  Loss of appetite - Related | 2 | 2 | 0
  Loss of appetite - Grade 3 related | 0 | 0 | 0
  Measles/Rubella-like rash - Any | 0 | 0 | 0
  Measles/Rubella-like rash - Grade 3 | 0 | 0 | 0
  Measles/Rubella-like rash - Related | 0 | 0 | 0
  Measles/Rubella-like rash - Grade 3 related | 0 | 0 | 0
  Fever - Any | 54 | 50 | 17
  Fever - Grade 3 | 3 | 2 | 2
  Fever - Related | 26 | 23 | 8
  Fever - Grade 3 related | 1 | 1 | 1

22. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) for All Groups, After Administration of Vitamin A and Study Vaccines at 6 Months of Age
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 30-day (Days 0-29) period after dose 1 of SB257049 and Vitamin A- Coad and RTS,S Groups, and 30-day period after Vitamin A administration - Control Group
Population: Analysis was performed on the Exposed set which included all subjects with first dose of the study vaccine + Vitamin A (Coad and RTS,S Groups) or Vitamin A (Control Group).
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 116 | 119 | 111

23. Secondary Outcome: Number of Subjects With Unsolicited AEs for the Coad Group and RTS,S Group, After Dose of Study Vaccines at 7.5 Months of Age
Description: as for outcome 22
Time Frame: Within 30-day (Day of vaccination and 29 subsequent days) period after dose 2 of SB257049 administered at Month 1.5 - Coad and RTS,S Groups
Population: Analysis was performed on the Exposed set which included all subjects with the second dose of the study vaccine administered (Coad and RTS,S Groups).
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 225 | 234
Participants | 107 | 109

24. Secondary Outcome: Number of Subjects With Unsolicited AEs for the Control Group, at Visit at 7.5 Months of Age
Description: as for outcome 22
Time Frame: During the 30-day period (Day of the visit and 29 subsequent days) after the visit at Month 1.5
Population: Analysis was performed on the Exposed set which included all subjects from the Control Group who completed the visit at Month 1.5.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 229
Participants | 80

25. Secondary Outcome: Number of Subjects With Unsolicited AEs for All Study Groups, After Dose of Study Vaccines Administered at 9 Months of Age
Description: as for outcome 22
Time Frame: Within 42-day (vaccination day and 41 subsequent days) period after dose 3 of SB257049 in Coad (+MeRu+YF vaccines) and RTS,S groups, and 42-day period after MeRU+YF vaccination in Control group, administered at Month 3
Population: Analysis was performed on the Exposed set which included all subjects with the third dose of the study vaccine for Coad (+MeRu+YF vacines) and RTS,S Groups, or MeRU + YF vaccine for the Control Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 222 | 231 | 227
Participants | 120 | 121 | 125

26. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs): All, Fatal and Related, for All Study Groups, Following Each Administration at Day 0, Month1.5 and Month 3
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During 30-Days period (Day of vaccination and 29 subsequent days) following each administration at Day 0, Month1.5 and Month 3 for Coad and RTS,S groups and at Day 0 and Month 3 in the Control Group.
Population: Analysis was performed on the Exposed set which included all subjects with at least one dose of the study vaccine or Vitamin A administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants
  Any SAEs | 13 | 8 | 16
  Fatal SAEs | 1 | 0 | 1
  Related SAEs | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects With Any SAEs for All Study Groups, From Day 0 Until Month 4.5
Description: as for outcome 26
Time Frame: From Day 0 up to Month 4.5
Population: Analysis was performed on the Exposed set which included all subjects with at least one dose of the study vaccines or Vitamin A administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 14 | 12 | 21

28. Secondary Outcome: Number of Subjects With Potential Immune-Mediated Disease (pIMDs) for All Study Groups From Day 0 Until Month 4.5
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurological disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 0 up to Month 4.5
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 0 | 0

29. Secondary Outcome: Number of Subjects With Meningitis for All Study Groups From Day 0 Until Month 4.5
Description: Meningitis is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It was assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to Month 4.5
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 0 | 0

30. Secondary Outcome: Number of Subjects With Seizures for All Groups, Post-vaccination for Vaccines Administered at 6, 7.5 or 9 Months of Age
Description: Seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It is assessed by the investigator as specific to the treatment administration.
Time Frame: Within 30 days post-vaccination for vaccine doses administered at Day 0, Month 1.5 or 42 days post-vaccination (doses given at Month 3 [Coad & Control Groups] or Month 4.5 [RTS,S Group]) vaccination period from Day 0 until Month 4.5
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 0 | 0

31. Secondary Outcome: Number of Subjects With Generalized Convulsive Seizure for All Study Groups, After Vaccines Administered at Day 0 and Month 1.5 (Coad and RTS,S Groups) and After Vaccines Administered at Month 3 (All Groups)
Description: Generalized convulsive seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It is assessed by the investigator as specific to the treatment administration.
Time Frame: Within 7 days after vaccines administered at Day 0 and Month 1.5 for the Coad and RTS,S groups and 14 days after vaccines administered at Month 3 for all groups
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 0 | 0

32. Secondary Outcome: Number of Subjects With Unsolicited AEs for the Coad Group and RTS,S Group, After the Booster Dose of Study Vaccine Administered at 27 Months of Age
Description: as for outcome 22
Time Frame: During the 30-day period (Day of vaccination and 29 subsequent days) after booster dose administered at Month 21
Population: Analysis was performed on the Exposed set which included all subjects with the booster dose of study vaccine administered at 27 months of age (Coad and RTS,S Groups)
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 216 | 209
Participants | 62 | 67

33. Secondary Outcome: Number of Subjects With Unsolicited AEs for the Control Group, After Dose of Study Vaccine Administered at 10.5, 11.5, 12.5 and 30 Months of Age
Description: as for outcome 22
Time Frame: During the 30-Day Period (Day of vaccination and 29 subsequent days) after primary doses of study vaccine administered at Month 4.5, Month 5.5, Month 6.5 (across primary doses), and after booster dose administered at Month 24
Population: Analysis was performed on the Exposed set which included all subjects with at least one dose of study vaccine administered at 10.5, 11.5, 12.5 and 30 months of age (Control Group).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 223
Participants
  Across primary doses | 160
  At Month 24: number analyzed (Participants) | 218
  At Month 24 | 57

34. Secondary Outcome: Number of Subjects With SAEs for All Study Groups From Day 0 Until Study End
Description: as for outcome 26
Time Frame: During the entire study period (From Day 0 until Month 33 for Coad and RTS,S Groups and Month 36 for the Control Group)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 61 | 62 | 66

35. Secondary Outcome: Number of Subjects With pIMDs for All Study Groups From Day 0 Until Study End
Description: as for outcome 28
Time Frame: During the entire study period (From Day 0 until Month 33 for Coad and RTS,S Groups and Month 36 for the Control Group)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 1 | 0

36. Secondary Outcome: Number of Subjects With Meningitis for All Study Groups From Day 0 Until Study End
Description: Meningitis is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It is assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (From Day 0 until Month 33 for Coad and RTS,S Groups and Month 36 for the Control Group)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group | Control Group
Number analyzed (Participants) | 231 | 236 | 232
Participants | 0 | 1 | 1

37. Secondary Outcome: Number of Subjects With Seizures for Vaccines Doses Administered at 6, 7.5, 27 Months of Age for Coad and RTS,S Groups; and at 9 Months of Age for Coad Group or 10.5 Months of Age for RTS,S Group
Description: Seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It was assessed by the investigator as specific to the treatment administration. Results are presented across all doses for Coad and RTS,S Groups.
Time Frame: Within 30 days post-vaccination (doses given at Day 0, Month 1.5, Month 21) & 42 days post-vaccination (dose given at Month 3 [Coad Group] or Month 4.5 [RTS,S Group])
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 231 | 236
Participants | 0 | 0

38. Primary Outcome: Anti-CS Antibody Concentrations, One Month Post Dose 3 of SB257049 (Study End Analysis)
Description: Concentrations were expressed as GMCs with the following unit of measure: EU/mL. The 95% confidence intervals were calculated using the ANOVA model. The antibody response of anti-CS was assessed in the Coad Group and the RTS,S Group. The analysis was re-evaluated and performed on the Per-Protocol set for immunogenicity defined at study end.
Time Frame: At one month post Dose 3 of SB257049 (Month 4)
Population: Analysis was performed on the Per-Protocol set for immunogenicity, defined at study end, which included all evaluable subjects meeting all eligibility criteria, complying with protocol defined procedures, with no elimination criteria during the study. Subjects with incomplete vaccination course or blood sampling performed outside protocol defined windows were eliminated. One subject that was eliminated at the primary analysis performed at Month 4.5 was included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Coad Group | RTS,S Group
Number analyzed (Participants) | 208 | 213
EU/mL | 454.51 [411.43 to 502.11] | 422.49 [382.89 to 466.18]
Statistical Analysis 1: Comparison: Coad Group vs RTS,S Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]

39. Secondary Outcome: Number of Subjects With Seizures for Vaccines Doses Administered at 10.5, 11.5, 12.5, 30 and 9 Months of Age for Control Group
Description: Seizure is an adverse event of specific interest (AESI). An AESI is defined as an AE including autoimmune diseases and other mediated inflammatory disorders. It was assessed by the investigator as specific to the treatment administration. Results are presented across all doses for the Control Group.
Time Frame: Within 30 days post-vaccination (doses given at Month 4.5, Month 5.5, Month 6.5, Month 24) & 42 days post-vaccination (dose given at Month 3)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 232
Participants | 1

ADVERSE EVENTS:
Time Frame: Solicited local & general AEs: Coad & RTS,S groups over 7-day follow-up period (FU) after vaccination at 6 & 7.5 Months of age (Mth-age); Control group at 6 Mth-age; all groups 14-Day FU after vaccination at 9 Mth-age. Unsolicited AEs: Coad & RTS,S groups over 30-Day FU after vaccination at 6, 7.5 & 27 Mth-age; Control group at 6, 10.5, 11.5, 12.5 & 30 Mth-age; all groups 42-Day FU after vaccination at 9 Mth-age. SAEs: Coad & RTS,S groups Day 0-Month 33; Control Group: Day 0-Month 36
Arm/Group | Coad Group | RTS,S Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/231 | 0/236 | 3/232
Serious Adverse Events (participants affected / at risk) | 61/231 | 62/236 | 66/232
Other Adverse Events (participants affected / at risk) | 219/231 | 221/236 | 207/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coad Group (N=231) | RTS,S Group (N=236) | Control Group (N=232)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 4 (4)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 3 (5) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Gastroenteritis (Infections and infestations) | 16 (16) | 17 (18) | 13 (13)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Malaria (Infections and infestations) | 6 (6) | 3 (3) | 11 (12)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 5 (5) | 4 (4)
Otitis media acute (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Plasmodium falciparum infection (Infections and infestations) | 21 (28) | 29 (35) | 21 (31)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (17) | 12 (14) | 17 (22)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Salmonella sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 2 (2) | 8 (8)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Exposure via ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coad Group (N=231) | RTS,S Group (N=236) | Control Group (N=232)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 17 (17) | 22 (28)
Enteritis (Gastrointestinal disorders) | 37 (42) | 42 (53) | 54 (77)
Infantile colic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 13 (14)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (5)
Injection site erythema (General disorders) | 11 (11) | 16 (16) | 2 (2)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 38 (38) | 31 (38) | 1 (1)
Injection site swelling (General disorders) | 15 (16) | 15 (15) | 1 (1)
Irritability postvaccinal (General disorders) | 31 (36) | 37 (43) | 6 (7)
Pyrexia (General disorders) | 101 (138) | 95 (133) | 28 (31)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 2 (2) | 3 (4) | 4 (4)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Body tinea (Infections and infestations) | 4 (4) | 5 (7) | 3 (3)
Bronchiolitis (Infections and infestations) | 5 (5) | 7 (7) | 5 (5)
Bullous impetigo (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 26 (27) | 25 (29) | 31 (34)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cutaneous larva migrans (Infections and infestations) | 8 (9) | 6 (6) | 7 (8)
Dermatitis infected (Infections and infestations) | 15 (16) | 23 (25) | 29 (37)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 12 (13) | 13 (13) | 15 (16)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Furuncle (Infections and infestations) | 14 (15) | 4 (5) | 9 (10)
Gastroenteritis (Infections and infestations) | 103 (139) | 120 (162) | 119 (192)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Helminthic infection (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 9 (10) | 4 (4) | 18 (20)
Injection site abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (2)
Malaria (Infections and infestations) | 44 (60) | 51 (65) | 76 (129)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Otitis media (Infections and infestations) | 20 (21) | 26 (28) | 30 (32)
Otitis media acute (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 40 (42) | 33 (37) | 30 (34)
Respiratory tract infection (Infections and infestations) | 67 (83) | 68 (88) | 84 (114)
Rhinitis (Infections and infestations) | 17 (17) | 20 (22) | 21 (22)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 16 (18) | 16 (17) | 25 (35)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tinea capitis (Infections and infestations) | 3 (4) | 1 (1) | 3 (3)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 143 (246) | 149 (239) | 168 (314)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3) | 4 (4)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 14 (14) | 6 (6) | 5 (5)
Viral rash (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 19 (20) | 24 (27) | 15 (15)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 17 (17) | 14 (15) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 23 (27) | 25 (28) | 28 (30)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02699099/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02699099/SAP_001.pdf